CLINICAL TRIAL: NCT03791190
Title: The Efficacy and Safety of Regional Citrate Anticoagulation Versus No-anticoagulation for CRRT in Patients With Liver Failure and High Risk Bleeding: a Randomized, Control, Open-labeled Clinical Trial
Brief Title: RCA for CRRT in Liver Failure and High Risk Bleeding Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Shiren sun, Professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RCA for CRRT in liver failure
Record Dates: First submitted 2018-11-12; First posted 2019-01-02 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-12

CONDITIONS: Liver Failure
Keywords: CRRT; liver failure; filter lifespan; bleeding
MeSH Terms: conditions — Liver Failure; Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No-anticoagulation (Active Comparator): Patients accepted no-anticoagulation CRRT. Blood flow 200 ml/h. The replacement fluid was infused 50% predilution and 50% post-dilution at the speed of 2 L/h.
  Interventions: Other: No-anticoagulation
- Regional citrate anticoagulation (Experimental): Patients accepted regional citrate anticoagulation. Blood flow 120-220 ml/h. Sodium citrate (4%) infusion before the filter in order to maintain post-filter ionCa2+ level between 0.25 to 0.35 mmol/L. Calcium gluconate supplementary after the filter to maintain serum ionCa2+ level between 1.0 to 1.2 mmol/L.
  Adjusting the infusion rate of sodium citrate and blood flow according to pre- and post-filtration ionCa2+.
  Adjusting the infusion rate of calcium gluconate according to the serum ionCa2+ level.
  Interventions: Other: Regional citrate anticoagulation

INTERVENTIONS:
Other: Regional citrate anticoagulation — Sodium citrate (4%) infusion before the filter in order to maintain post-filter ionCa2+ level between 0.25 to 0.35 mmol/L. Calcium gluconate supplementary after the filter to maintain serum ionCa2+ level between 1.0 to 1.2 mmol/L.
  Other Names: RCA
  Arms: Regional citrate anticoagulation
Other: No-anticoagulation — Patients accepted CRRT without anticoagulant.
  Arms: No-anticoagulation

SUMMARY:
The purpose of this single center, randomized, control, open-labeled study is to evaluate the effect and safety of RCA versus no anticoagulation for CRRT in patients with liver failure and high risk bleeding.

DETAILED DESCRIPTION:
Liver failure (LF) is a common co-morbidity in critical care patients who need continuous renal replacement therapy (CRRT). Patients with LF are usually associated with impaired coagulation, impaired metabolic ability of anticoagulants, and increased bleeding risk. KDIGO guideline recommended no-anticoagulation for CRRT in patients with liver failure and increased bleeding risk. However, the averaged CRRT circuit lifespan under no-coagulation was reported to be 7-8 hours in patients with liver failure. Commonly, a CRRT regimen needs more than 24 hours treatment, which means 3-4 filters replacement for one regimen in liver failure patients underwent no-anticoagulation CRRT. Several observational studies suggested that regional citrate anticoagulation (RCA) during CRRT was effective and safe in patients with liver failure. Therefore, the current opinions on the anticoagulation strategy for CRRT in patients with liver failure and high bleeding risk are controversial. Therefore, the purpose of this single center, randomized, control, open-labeled study is to evaluate the effect and safety of RCA versus no anticoagulation for CRRT in patients with liver failure and high risk bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Liver failure (acute liver failure and chronic liver failure)
* High bleeding risk
* Scheduled CRRT treatment
* Informed consent

Exclusion Criteria:

* Use of other anticoagulants
* Uncorrectable hypoxemia (PaO2 < 60 mmHg) or systemic hypoperfusion shock
* Pregnancy or lactation
* Fistula, CRRT treatment time < 12 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-09-06 (Actual); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
Filter failure | 72 hours
  Filter failure

SECONDARY OUTCOMES:
Serum Total Ca2+/ion Ca2+ level | 2, 6, 12, 20, 28, 36, 44, 52, 60, and 72 hours.
  Serum Total Ca2+/ ionized Ca2+ level
Hypocalcemia | 72 hours
  Ionized Ca2+ < 1.0
Acidosis | 72 hours
  Blood pH < 7.35
Alkalosis | 72 hours.
  Blood pH > 7.45
Bleeding | 72 hours
  Bleeding episode during the CRRT.
Serum citrate concentration | 2, 6, 12, 20, 28, 36, 44, 52, 60, and 72 hours.
  Citrate concentration
Serum total bilirubin level | Every 24 hours up to 72 hours.
  Total bilirubin
Serum AST level | Every 24 hours up to 72 hours.
  AST
Serum ALT level | Every 24 hours up to 72 hours.
  ALT

CONTACTS AND LOCATIONS:
Overall Officials: Shiren Sun, Doctor, Study Chair — Xijing Hospital, the Fourth Military Medical University; Ming Bai, Doctor, Principal Investigator — Xijing Hospital, the Fourth Military Medical University
Locations (1):
- Xijing Hospital of Nephrology, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Bai M, Yu Y, Zhao L, Tian X, Zhou M, Jiao J, Liu Y, Li Y, Yue Y, Wei L, Jing R, Li Y, Ma F, Liang Y, Sun S. Regional Citrate Anticoagulation versus No Anticoagulation for CKRT in Patients with Liver Failure with Increased Bleeding Risk. Clin J Am Soc Nephrol. 2024 Feb 1;19(2):151-160. doi: 10.2215/CJN.0000000000000351. Epub 2023 Nov 6. PMID 37990929